CLINICAL TRIAL: NCT05447026
Title: The Adjunctive Use of Antimicrobial Photodynamic Therapy, Light-emitting-diode Photobiomodulation, and Ozone Therapy in Regenerative Treatment of Stage III Grade C Periodontitis
Brief Title: The Effect of Adjunctive Therapies in Regenerative Treatment of Stage III Grade C Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/105
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis; Lasers; Ozone; Wound Healing; Regeneration
MeSH Terms: conditions — Periodontitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The present study is a parallel design randomized controlled clinical trial evaluating four different treatment approaches.
Who Masked: Investigator
Masking Description: An examiner, who was blinded for the patient group assignment, performed clinical measurements, and sample collections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Active Comparator): Regenerative surgical treatment of periodontal infrabony defects without any adjunctive therapies.
  Interventions: Device: Control group
- antimicrobial photodynamic therapy (aPDT) group (Active Comparator): Regenerative surgical treatment of periodontal infrabony defects in conjunction with irradiation by a diode laser and a photosensitizer
  Interventions: Device: Antimicrobial photodynamic therapy (aPDT) group
- LED photobiomodulation group (Active Comparator): Regenerative surgical treatment of periodontal infrabony defects in conjunction with irradiation by a LED device
  Interventions: Device: LED photobiomodulation group
- Topical ozone group (Active Comparator): Regenerative surgical treatment of periodontal infrabony defects in conjunction with topical ozone application
  Interventions: Device: Topical ozone group

INTERVENTIONS:
Device: Control group — Following local anesthesia, a full-thickness (muco-periosteal) access flap was elevated, granulation tissue was removed and direct instrumentation of the affected root surfaces was performed under the saline irrigation. Intrabony defects were filled with granules of allograft bone material and covered with a native porcine pericardial collagen membrane. The flaps were repositioned and sutured without any tension in order to achieve primary closure of the inter-dental area using a 5-0 mono-filament non-resorbable PTEF suturing material. On the 1st, 3rd, and 7th postoperative days, the sites in the control group received only saline irrigation for 1 min.
  Arms: Control group
Device: Antimicrobial photodynamic therapy (aPDT) group — Following local anesthesia, a full-thickness (muco-periosteal) access flap was elevated, granulation tissue was removed and direct instrumentation of the affected root surfaces was performed under the saline irrigation. Intrabony defects were filled with granules of allograft bone material and covered with a native porcine pericardial collagen membrane. The flaps were repositioned and sutured without any tension in order to achieve primary closure of the inter-dental area using a 5-0 mono-filament non-resorbable PTEF suturing material. On the 1st, 3rd, and 7th postoperative days, aPDT group received additional application of a diode laser with a wavelength of 810 nm and a power rating of 200 mW (continuous mode). Indocyanine-green (ICG) as a photosensitizer at a concentration of 1 mg/ml was applied at the surgical site on both the buccal and the lingual sides of the flaps. Irradiation was performed in non-contact mode in a constant distance of 1 mm during 30 s per site
  Arms: antimicrobial photodynamic therapy (aPDT) group
Device: LED photobiomodulation group — Following local anesthesia, a full-thickness (muco-periosteal) access flap was elevated, granulation tissue was removed and direct instrumentation of the affected root surfaces was performed under the saline irrigation. Intrabony defects were filled with granules of allograft bone material and covered with a native porcine pericardial collagen membrane. The flaps were repositioned and sutured without any tension in order to achieve primary closure of the inter-dental area using a 5-0 mono-filament non-resorbable PTEF suturing material. On the 1st, 3rd, and 7th postoperative days, irradiation was carried out with a LED device with a wavelength of 626 nm in the near-infrared region at a dose of 20 mw/cm2 for 20 min with a total energy of 222 J
  Arms: LED photobiomodulation group
Device: Topical ozone group — Following local anesthesia, a full-thickness (muco-periosteal) access flap was elevated, granulation tissue was removed and direct instrumentation of the affected root surfaces was performed under the saline irrigation. Intrabony defects were filled with granules of allograft bone material and covered with a native porcine pericardial collagen membrane. The flaps were repositioned and sutured without any tension in order to achieve primary closure of the inter-dental area using a 5-0 mono-filament non-resorbable PTEF suturing material. On the 1st, 3rd, and 7th postoperative days, topical ozone group received ozone application with an ozone generator at 80% concentration using probe #3 for 30 s per site
  Arms: Topical ozone group

SUMMARY:
Anti-infective procedures play a very important role in the success of regenerative surgical treatment of aggressive periodontitis, Grade C periodontitis, which shows the newly named molar-incisor pattern according to the 2017 World Workshop Classification of Periodontal Diseases. In the present study, it was aimed to analyze the effects of photodynamic, photobiomodulation, and ozone therapy applications on periodontal healing, both clinically and immunologically, in addition to the surgical regenerative treatment of aggressive periodontitis. Forty adult individuals diagnosed with aggressive periodontitis who applied to Gazi University Faculty of Dentistry Department of Periodontology for the treatment of periodontal disease were included in the study. In addition to the regenerative surgical treatment using cortico-cancellous particle allograft and a resorbable collagen membrane in randomly determined areas with multiple intraosseous defects, topical ozone, antimicrobial photodynamic, and light-emitting diode (LED) photobiomodulation treatments were applied. Periodontal clinical parameters [plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing pocket depths (PPD), clinical attachment level (CAL), gingival recession (GR), and width of keratinized gingival (WKG)] were examined and patient-centered postoperative evaluations, and early wound healing index (EHI) assessments were performed for 2 weeks after the operation. In addition, gingival crevicular fluid (GCF) samples from patients to determine the total amount and concentration of vascular endothelial growth factor (VEGF), interleukin -6 (IL-6), Runt-related transcription factor 2 (RunX2), NEL-like 1 (Nell-1), Osterix and samples were quantified by Quantitative Real-Time PCR. The repeated measures ANOVA model was used for the analysis of variables in which both group and time measurements were taken.

DETAILED DESCRIPTION:
Periodontitis is a chronic multifactorial inflammatory disease driven by the dysbiotic relationship between the host immune-inflammatory response and the commensal oral microbiota in plaque biofilms that results in the progressive destruction of the tooth-supporting apparatus (Papapanou et al., 2018). Several modifiable and non-modifiable factors including genetic, environmental, and systemic factors can influence its pathogenicity and alter patient's susceptibility to the development and severity of the periodontal disease (Kinane et al., 2017).

According to the 2017 World Workshop classification, stages III or IV, grade C periodontitis, formerly defined as aggressive periodontitis, is characterized by the rapid progression of a particularly severe form of periodontal disease (Papapanou et al., 2018). According to the EFP S3 Clinical Treatment Guidelines, in patients with deep periodontal pockets (≥ 6 mm) step 2 of periodontal therapy (subgingival instrumentation, with or without adjunctive therapies) may be insufficient, and step 3 of surgical periodontal therapy incorporated with regenerative procedures may be required to eliminate deep residual pockets and reconstruct the intrabony part of the defects, as well as prevent tooth loss (Sanz et al., 2020). Despite of some limitations of access flap periodontal surgeries such as increased risk of gingival recession, increased postoperative dentin hypersensitivity, and morbidity, regenerative surgical procedures have been shown to be efficacious for the treatment of intrabony defects in patients with severe periodontitis, with the rapid rate of progression (Diaz-Faes et al., 2020). To improve the outcomes of therapy in severe periodontitis patients, adjunctive interventions such as local or systemic antibiotics, and antimicrobial photodynamic or photobiomodulation therapies using lasers or light-emitting-diodes (LED) have been explored in non-surgical and surgical treatment approaches (Collins et al., 2022; Andere et al., 2022; Giannelli et al., 2018).

Within the visible red or near-infrared (NIR) range of the spectrum (600 to 700 nm and 780 to 1100 nm), low-level lasers (LLL) or LEDs have been widely utilized as an adjunct therapy for periodontitis treatment based on their photobiomodulation and decontamination effects, which primarily occur at the level of the cellular respiratory chain (Zhao et al., 2021). These modalities promote mitochondrial activity and activate the mechanisms, i.e., inducing intracellular metabolic changes, enhancing the cellular resuscitation system, increasing adenosine triphosphate (ATP) and extracellular matrix (ECM) production (Heidari et al., 2018). Through the biological characteristics of these approaches, various studies have shown to increase angiogenesis, promote modulation of the immunoinflammatory response, stimulate the processes of regeneration and epithelialization, and reduce postoperative symptoms. The use of LLLs or LEDs in conjunction with photosensitizing agents (optical absorption-dye) has been referred as antimicrobial photodynamic therapy (aPDT). This procedure stimulates the dye to form free radicals of singlet oxygen that will act as toxic to the target cells or bacteria mainly as a result of deterioration to the cytoplasmic membrane and DNA, thereby demonstrating anti-microbial activity at periodontal pathogenic bacteria in combination with periodontal treatment (Katsikanis et al., 2020). Similar to the biostimulatory features of LLLs or LEDs, adjunctive gaseous ozone therapy applications have been recently exploited because of their analgesic, immunomodulatory, and anti-inflammatory effects, which may have the ability to provide significant added benefits in both step 2 and 3 of the periodontal therapy due to its analgesic, immunomodulatory, and anti-inflammatory effects (Rapone et al., 2022). All these adjunct therapies have also been shown to have a positive effect on the proliferation and osteogenic differentiation of undifferentiated periodontal tissue cells or the direct stimulation of osteoblasts in several studies. However, little information exists regarding the efficacy of these modalities adjunct to the periodontal regenerative therapies on the processes and sequences of the healing and consequently, in the postoperative expression levels of biomarkers of inflammation, angiogenesis, and osteogenesis. Therefore, the objectives of the present study were: (i) to investigate the additional influence of multiple sessions of aPDT, LED photobiomodulation, and topical gaseous ozone therapy applications associated with surgical regenerative treatments by using an allogenic bone graft in combination with a collagen membrane on clinical and patient-centered outcomes in patients with stage III, grade C periodontitis, and (ii) to analyze mRNA expression levels of vascular endothelial growth factor (VEGF), interleukin -6 (IL-6), runt-related transcription factor 2 (RunX2), NEL-like 1 (Nell-1), and osterix in gingival crevicular (GCF) samples at baseline and the 1-, 3- and 6-month follow-ups after the treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

* the presence of ≥ 20 teeth (excluding third molars);
* the presence of infrabony defects of ≥ 3 mm as detected in periapical radiographs;
* have not received any periodontal treatment and have not taken any of antibiotics within the last 6 months.

Exclusion Criteria:

* females that were pregnant or breastfeeding;
* systemic disease that could affect the risk or progression of periodontal disease (e.g., diabetes mellitus, bone metabolic disease, blood disorders, radiation or immuno-suppressive therapy);
* medications that significantly impact periodontal inflammation and bone metabolism (nonsteroidal anti-inflammatory drugs, bisphosphonates, selective serotonin reuptake inhibitors [SSRIs], proton pump inhibitors [PPIs], calcium channel blockers (CCBs), benzodiazepines, or corticosteroids);
* smokers or use of other tobacco products;
* teeth with class III furcation lesions or mobility degree >1;
* systemic antimicrobial treatment (up to 3 weeks prior study inclusion);
* periodontal treatment within the past 6 months prior to recruitment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in CAL values | 6 months after the surgery
  The changes in the mean CAL values between baseline and postoperative 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Ozbay, Prof Dr, Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Result] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Result] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Result] Diaz-Faes L, Fernandez-Somoano A, Magan-Fernandez A, Mesa F. Efficacy of regenerative therapy in aggressive periodontitis: a systematic review and meta-analysis of randomised controlled clinical trials. Clin Oral Investig. 2020 Apr;24(4):1369-1378. doi: 10.1007/s00784-020-03237-0. Epub 2020 Feb 14. PMID 32060656
- [Result] Collins JR, Ogando G, Gonzalez R, Figuero E, Marin MJ, Sanz M, Herrera D. Adjunctive efficacy of systemic metronidazole in the surgical treatment of periodontitis: a double-blind parallel randomized clinical trial. Clin Oral Investig. 2022 May;26(5):4195-4207. doi: 10.1007/s00784-022-04392-2. Epub 2022 Feb 5. PMID 35122549
- [Result] Andere NMRB, Castro Dos Santos NC, Araujo CF, Paz HES, Shaddox LM, Casarin RCV, Santamaria MP. Open flap debridement compared to repeated applications of photodynamic therapy in the treatment of residual pockets: A randomized clinical trial. J Periodontol. 2022 Nov;93(11):1671-1681. doi: 10.1002/JPER.22-0059. Epub 2022 Jun 2. PMID 35536044
- [Result] Giannelli M, Materassi F, Fossi T, Lorenzini L, Bani D. Treatment of severe periodontitis with a laser and light-emitting diode (LED) procedure adjunctive to scaling and root planing: a double-blind, randomized, single-center, split-mouth clinical trial investigating its efficacy and patient-reported outcomes at 1 year. Lasers Med Sci. 2018 Jul;33(5):991-1002. doi: 10.1007/s10103-018-2441-9. Epub 2018 Jan 18. PMID 29349511
- [Result] Zhao H, Hu J, Zhao L. The effect of low-level laser therapy as an adjunct to periodontal surgery in the management of postoperative pain and wound healing: a systematic review and meta-analysis. Lasers Med Sci. 2021 Feb;36(1):175-187. doi: 10.1007/s10103-020-03072-5. Epub 2020 Jul 1. PMID 32613416
- [Result] Heidari M, Fekrazad R, Sobouti F, Moharrami M, Azizi S, Nokhbatolfoghahaei H, Khatami M. Evaluating the effect of photobiomodulation with a 940-nm diode laser on post-operative pain in periodontal flap surgery. Lasers Med Sci. 2018 Nov;33(8):1639-1645. doi: 10.1007/s10103-018-2492-y. Epub 2018 Jul 6. PMID 29978268
- [Result] Katsikanis F, Strakas D, Vouros I. The application of antimicrobial photodynamic therapy (aPDT, 670 nm) and diode laser (940 nm) as adjunctive approach in the conventional cause-related treatment of chronic periodontal disease: a randomized controlled split-mouth clinical trial. Clin Oral Investig. 2020 May;24(5):1821-1827. doi: 10.1007/s00784-019-03045-1. Epub 2019 Aug 13. PMID 31410672
- [Result] Rapone B, Ferrara E, Santacroce L, Topi S, Gnoni A, Dipalma G, Mancini A, Di Domenico M, Tartaglia GM, Scarano A, Inchingolo F. The Gaseous Ozone Therapy as a Promising Antiseptic Adjuvant of Periodontal Treatment: A Randomized Controlled Clinical Trial. Int J Environ Res Public Health. 2022 Jan 16;19(2):985. doi: 10.3390/ijerph19020985. PMID 35055807